CLINICAL TRIAL: NCT03595098
Title: Treatment Effects of Family Based Cognitive Therapy in Children and Adolescents With Obsessive Compulsive Disorder
Acronym: TECTO
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Anne Katrine Pagsberg (Other)
Collaborators: Danish Research Centre for Magnetic Resonance (Other); Copenhagen Trial Unit, Center for Clinical Intervention Research (Other)
Responsible Party: Sponsor-Investigator, Anne Katrine Pagsberg, Associate professor at Child and Adolescent Mental Health Centre, Copenhagen, Copenhagen Trial Unit, Center for Clinical Intervention Research
Organization: Copenhagen Trial Unit, Center for Clinical Intervention Research (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TECTO
Record Dates: First submitted 2018-05-03; First posted 2018-07-23 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-07

CONDITIONS: Obsessive-Compulsive Disorder in Children; Obsessive-Compulsive Disorder in Adolescence
Keywords: OCD
MeSH Terms: interventions — Relaxation Therapy

STUDY DESIGN:
Intervention Model Description: single-centre, parallel group superiority randomised clinical trial with blinded outcome assessment
Who Masked: Outcomes Assessor
Masking Description: Due to the nature of the interventions, it is not possible to blind the participants, the investigators administrating the interventions (therapists, i.e. medical doctors and clinical psychologists, and other caregivers), or parents. Blinding will be applied in all possible aspects of the trial such as: outcome assessment and MRI-scanning and neuropsychological testing. Additionally data managers, statisticians, and investigators drawing conclusions, will be fully blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FCBT (Experimental): The Family Based Cognitive Behavioural Therapy (FCBT)
  Interventions: Behavioral: Family Based Cognitive Behavioural Therapy
- FPRT (Active Comparator): Family-based Psychoeducation /Relaxation Training (FPRT)
  Interventions: Behavioral: Family Based Psychoeducation/Relaxation Training

INTERVENTIONS:
Behavioral: Family Based Cognitive Behavioural Therapy — Family Based Cognitive Behavioural Therapy (FCBT) focuses on the interrelation between thought, emotion, and behaviour, Exposure and Response Prevention, family involvement, homework assignments, and formulating of specific goals for the child. The important, active components is Exposure and Response Prevention. It involves exposing the child to a feared object, situation or thought, and preventing the child from carrying out compulsions to show the child that distress/anxiety can decrease or disappear without performing rituals.
  Arms: FCBT
Behavioral: Family Based Psychoeducation/Relaxation Training — Family-based Psychoeducation/Relaxation Training (FPRT) as an active control matches the experimental intervention as closely as possible, many elements of the control intervention are similar to FCBT. The main and intended difference between the two approaches is the absence of the Exposure and Response Prevention component, which is deemed the most effective treatment for OCD.
  Arms: FPRT

SUMMARY:
To investigate the benefits and harms, and the neural and neurocognitive mediators of treatment response, in family-based cognitive behavioural therapy versus family-based psychoeducation and relaxation training in children and adolescents with obsessive compulsive disorder. The aim is to conduct this investigation in an optimal trial design with the lowest possible risk of bias.

DETAILED DESCRIPTION:
Obsessive-compulsive disorder is the fourth most common psychiatric disorder, affecting 1-3% of children and adolescents globally. The recommended first-line treatment is cognitive behavioral therapy with exposure and response prevention. Yet, more than 40% of patients do not, or only partially, benefit from therapy. A better understanding of the mechanisms underlying response to cognitive behavioral therapy is needed to improve treatment. In the TECTO study, we will conduct a combined randomized clinical trial and longitudinal case-control study to elucidate how neural, cognitive, emotional, and neuroendocrine factors moderate and mediate treatment response. At baseline, 128 children and adolescents with obsessive-compulsive disorder will be compared to 128 healthy control participants to map neurobiological, cognitive, and emotional markers of obsessive-compulsive disorder. After baseline assessment, patients are randomly assigned to 16 weeks of either cognitive behavioral therapy with exposure and response prevention or an active control treatment with psychoeducation and relaxation training. This design allows us to test how factors that are specific to cognitive behavioral therapy (e.g. exposure and response prevention) contribute to observed treatment effects. Our primary outcome is OCD symptom severity measured with the Children's Yale-Brown Obessive-Compulsive Scale. Secondary outcomes are health-related quality of life and negative treatment effects. To detect neural and cognitive mediators of treatment, we will measure brain structure and function, and cognitive performance, at baseline and end-of-treatment. Furthermore, we will monitor a range of therapeutic, emotional, family, and neuroendocrine factors before, during, and after treatment. We expect that findings from TECTO will have important theoretical implications and will help refine our understanding of OCD as a heterogeneous and multidimensional disorder. Finally, we expect that our findings will contribute significantly to the improvement of psychotherapy and development of more targeted interventions for pediatric obsessive-compulsive disorder, which can minimize the use of medication, prevent chronicity, and reduce the substantial socioeconomic burden of the disorder.

ELIGIBILITY:
Inclusion Criteria:

* OCD diagnosis as primary diagnosis, meeting the criteria for International Classification of Diseases 10 (ICD-10) F42, verified with a semi-structured psychopathological interview using Schedule for Affective Disorders and Schizophrenia for school-aged children, Present and Lifetime version (K-SADS-PL).
* Children's Yale-Brown Obsessive-Compulsive Scale (CY-BOCS) entry score ≥16, a cut-off score used in previous studies.
* Age 8 through 17 years (both inclusive).
* Signed informed consent.

Exclusion Criteria:

* Comorbid illness that contraindicates trial participation: pervasive developmental disorder not including Asperger's syndrome (ICD-10 F84.0-84.4 + F84.8-84.9), schizophrenia/paranoid psychosis (ICD-10 F20-25 + F28-29), mania or bipolar disorder (ICD-10 F30 and F31), depressive psychotic disorders (F32.3 + F33.3), substance dependence syndrome (ICD-10 F1x.2).
* Intelligence Quotient <70.
* Treatment with Cognitive Behavioural Therapy (CBT), Serotonin Reuptake Inhibitors, or other antidepressant medication or antipsychotic medication within the last 6 months prior to trial entry.
* For MRI-scanning:

  * metal braces on teeth or metal implants;
  * any known brain pathology;
  * history of severe head-trauma (ICD-10 S6-S9);
  * pregnancy.

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 128 (Estimated)
Dates: Start 2018-08-28 (Actual); Primary Completion 2022-04-07 (Actual); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Children's Yale-Brown Obsessive-Compulsive Scale (CY-BOCS) score | Week 0, 4, 8, 16 and 40
  Children's Yale-Brown Obsessive-Compulsive Scale (CY-BOCS) is a 10-item questionnaire assessing the severity of obsessive compulsive disorder (OCD). Severity of compulsions and obsessions are rated on a scale from 0 (none) to 4 (extreme). The total score is calculated by summing the 10 individual scores and ranges from 0 to 40, where higher scores indicate more extreme symptoms.

SECONDARY OUTCOMES:
health-related quality of life assesses with KIDSCREEN-52 | Week 0, 4, 8, 16 and 40
  The KIDSCREEN instruments assess children's and adolescents' subjective health and well-being- health-related quality of life (HRQoL). Questionnaire consisted of 52 items which assessed HRQoL in 10 dimensions: physical well-being, psychological well-being, moods and emotions, self perception, autonomy, relation with parents and home life, social support and peers, school environment, social acceptance, and financial resources. Rasch scores are computed for each dimension and are transformed into T-values with a mean of 50 and a standard deviation of 10; higher scores indicate better HRQoL and well-being.
Occurrence of negative adverse events | Week 4, 8, 16 and 40
  The occurrence of negative adverse events is assessed with the Negative Effects Questionnaire (NEQ). The questionnaire is used for both parental reports and self-reports. It consists of 32 items that are scored on a five-point Likert-scale (0-4) where the highest value represents a severe negative effect of the event. The questionnaire differentiates between negative effects that are attributed to the treatment and those possibly caused by other circumstances, as well as one open-ended question.

OTHER OUTCOMES:
Magnetic resonance imaging | Week 0 and 16
  This is exploratory outcome. Magnetic resonance imaging (MRI) is used to obtain images of the patients' brains before and after treatment and the scanning consists of both structural and functional scans. From the functional scans response-inhibition-related and switch-related activity during Stop Signal Task performance and Task Switching performance is examined.
Family Accommodation Scale | Week 4, 8, 16 and 40
  This is exploratory outcome showing family factors. Family Accommodation Scale (FAS): a 13-item parent-report measure designed to assess accommodation of a child's OCD-related behaviors over the previous month. In an effort to assess multiple dimensions to accommodations (rather than one in isolation), items are anchored with respect to either frequency or magnitude utilizing a 5-pt Likert scale ranging from 0 (Never) to 4 (Daily) with higher scores indicating greater parental accommodation.
Family Environment Scale | Week 0
  This is exploratory outcome showing family factors. Family Environment Scale (FES)is composed of 90 items and 10 subscales that measure actual, preferred, and expected family social environments. The 10 subscales assess three dimensions: relationship dimensions, personal growth (or goal orientation) dimensions, and system maintenance dimensions. There are three FES forms (real, ideal, and expectations); only the FES real form will be used, which examines a family member's perception of the family as it is. The scale ranges from 10 to 40, with a score of 10 being representative of no family conflict and a score of 40 being representative of the greatest magnitude of family conflict. Therefore, a decrease in score represents a decrease in self-reported family conflict.
Parental Stress Scale | Week 4, 8, 16 and 40
  This is exploratory outcome showing family factors. Parental Stress Scale (PSS)measures parental stress in the parental relationship and consists of 18 items. The parent answers different statements about his or her relationship to the child by scoring each item on a five-point Likert-scale (1-5), 5 representing the highest amount of agreement with the statement and 1 representing the highest amount of dis-agreement. The positively formulated items are scored in reverse. PSS is thus scored on a scale from 18 to 90, where higher scores reflect greater stress.
Child Obsessive-Compulsive Impact Scale | Week 4, 8, 16 and 40
  This is exploratory clinical outcome.Child Obsessive-Compulsive Impact Scale (COIS) is a 33-item parent-report and self-report questionnaire that assesses OCD-related impairment in various areas of the child's life, including school, social, and home/family activities. For each item, the respondent rates the child's level of impairment on a 4-point Likert scale from 0 (not at all) to 3 (very much). The total score (0-99) is the sum of the item scores. Higher scores reflect more severe impairment.
Clinical Global Impression Severity and Clinical Global Impression Improvement Scale | Week 4, 8, 16 and 40
  This is exploratory clinical outcome. Clinical Global Impression Severity and Clinical Global Impression Improvement Scale (CGI-I and CGI-S) measure symptom severity, treatment response, and the efficacy of treatments in treatment studies of patients with mental disorders. Therefore higher scores indicate a worse mental state of the patient. The CGI is rated on a 7-point scale, with the severity of illness scale using a range of responses from 1 (normal) through to 7 (amongst the most severely ill patients). CGI-I scores range from 1 (very much improved) through to 7 (very much worse).
Occurrence of Serious Adverse Events | Week 0-Week 40
  This is exploratory clinical outcome. Occurrence of Serious Adverse Events.Any adverse events such as results in death, is life-threatening, requires hospitalisation or prolongs existing hospitalisation, results in persistent or significant disability or incapacity, or is a congenital anomaly or birth defect, which does not necessarily have a causal relationship with the intervention will be registered register.
Children's Global Assessment Scale | Week 4, 8, 16 and 40
  This is exploratory clinical outcome. Children's Global Assessment Scale Scale is a numeric scale used by mental health clinicians to rate the general functioning of youths under the age of 18. It is the 100-point single-item score, scored from 0-100 (worse to normal).
Remission | Week 16
  This is exploratory clinical outcome. Proportion of patients no longer meeting the diagnostic criteria for OCD, ICD-10 F.42 assessed with Schedule for Affective Disorders and Schizophrenia for school-aged children, Present and Lifetime version (K-SADS-PL) at the end of the intervention (remission).
OCD symptoms remission | Week 16
  This is exploratory clinical outcome.This is a binary, exploratory, clinical outcome. Treatment response based on the definition of a reduction in CY-BOCS score at week 16 of at least 30% in intraindividual comparison with the score at week 0.
Toronto Obsessive-Compulsive Rating Scale | Week 0 and week 16
  This is an exploratory clinical outcome. Toronto Obsessive-Compulsive Rating Scale (TOCS) is a quantitative and multidimensional measure of Obsessive-Compulsive traits in children and adolescents. Questionnaire with 21 items, and each item is scored on a 7-point likert scale from -3 to 3. Dimension scores ranges from -3 to 3. The total scale ranges from -63 to 63. Higher values represents worse outcome.
Risk taking and decision-making ability | Week 0 and week 16th
  This is exploratory cognition outcome. Risk taking and decision-making assessed by Cambridge Gambling Task
Planning ability | Week 0 and week 16th
  This is exploratory cognition outcome. Planning ability assessed by Stockings of Cambridge test. It is a computerized neuropsychological test assessing executive functions. There are two main outcomes: Reaction time and accuracy. Low reaction time combined with high accuracy represents better planning ability.
Working memory capacity | Week 0 and week 16th
  This is exploratory cognition outcome. Working memory capacity assessed by Spatial Working Memory test. It requires retention and manipulation of visuospatial information. This self-ordered test has notable executive function demands and provides a measure of strategy as well as working memory errors. Reaction time and accuracy. Low reaction time combined with high accuracy represents better memory capacity.
Motor skills | Week 0 and week 16th
  This is an exploratory cognition outcome. Motor skills assessed with Purdue Pegboard test. It controls for potential effects of differences in motor skills on performance on other tasks in the battery. Test is a rectangular board with 2 sets of 25 holes running vertically and 4 concave cups at the top. Small metal pegs are placed in the cup on the side being tested, with subjects asked to remove the pegs and place them vertically in the holes as rapidly as possible. The number of pegs placed in 30 seconds is scored. More accurate placed pegs represent better motor skills.
Habit formation | Week 0 and week 16th
  This is exploratory cognition outcome. Weather Prediction Learning Task, which is a probabilistic classification learning task in which participants learn to predict the weather (i.e. "sun" or "rain" outcomes) based on combinations of cues that predict "sun" versus "rain" outcomes. Better prediction mean better outcome.
Change in Delis-Kaplan Executive Function System (D-KEFS) | Week 0 and week 16th
  This is an exploratory cognition outcome.The Delis-Kaplan Executive Function System (DKEFS). Test three tests from D-KEFS will be used: Trail Making, Verbal Fluency, and Design Fluency. The three test measures set-shifting ability, processing speed, and response inhibition. Each test has a scaled score going from 1-19, where higher values represent better outcome.
Change in Thought-Action Fusion Questionnaire for Adolescents | Week 0, 4, 8, 16 and 40
  This is exploratory outcome. Thought-Action Fusion Questionnaire for Adolescents (TAFQ-A): a 15-item questionnaire measuring cognitive biases that are thought to play an important role in the development of obsessions. Each item is scored on a 4-point likert scale from 1-4, were higher values represent worse outcome.
Executive function | Week 0 and week 16
  This is exploratory outcome. Behaviour Rating Inventory of Executive Function: a self-report and parent-report questionnaire assessing impairment of executive function. Executive function in daily life (range:70-210). Higher score indicate greater executive dysfunction.

CONTACTS AND LOCATIONS:
Overall Officials: Anne Katrine Pagsberg, Professor, Principal Investigator — Child and Adolescent Mental Health Centre, Copenhagen
Locations (1):
- Child and Adolescent Mental Health Centre, Bispebjerg, Copenhagen, Denmark

REFERENCES:
- [Derived] Pretzmann L, Christensen SH, Bryde Christensen A, Funch Uhre C, Uhre V, Thoustrup CL, Clemmesen IT, Gudmandsen TA, Korsbjerg NLJ, Mora-Jensen AC, Ritter M, Olsen MH, Clemmensen LKH, Lindschou J, Gluud C, Thomsen PH, Vangkilde S, Hagstrom J, Rozental A, Jeppesen P, Verhulst F, Hybel KA, Lonfeldt NN, Plessen KJ, Poulsen S, Pagsberg AK. Adverse events in cognitive behavioral therapy and relaxation training for children and adolescents with obsessive-compulsive disorder: A mixed methods study and analysis plan for the TECTO trial. Contemp Clin Trials Commun. 2023 Jun 20;34:101173. doi: 10.1016/j.conctc.2023.101173. eCollection 2023 Aug. PMID 37497354
- [Derived] Olsen MH, Hagstrom J, Lonfeldt NN, Uhre C, Uhre V, Pretzmann L, Christensen SH, Thoustrup C, Korsbjerg NLJ, Mora-Jensen AC, Ritter M, Engstrom J, Lindschou J, Siebner HR, Verhulst F, Jeppesen P, Jepsen JRM, Vangkilde S, Thomsen PH, Hybel K, Clemmesen LKH, Gluud C, Plessen KJ, Pagsberg AK, Jakobsen JC. Family-based cognitive behavioural therapy versus family-based relaxation therapy for obsessive-compulsive disorder in children and adolescents (the TECTO trial): a statistical analysis plan for the randomised clinical trial. Trials. 2022 Oct 6;23(1):854. doi: 10.1186/s13063-022-06799-4. PMID 36203215
- [Derived] Pagsberg AK, Uhre C, Uhre V, Pretzmann L, Christensen SH, Thoustrup C, Clemmesen I, Gudmandsen AA, Korsbjerg NLJ, Mora-Jensen AC, Ritter M, Thorsen ED, Halberg KSV, Bugge B, Staal N, Ingstrup HK, Moltke BB, Kloster AM, Zoega PJ, Mikkelsen MS, Harboe GS, Larsen KF, Clemmensen LKH, Lindschou J, Jakobsen JC, Engstrom J, Gluud C, Siebner HR, Thomsen PH, Hybel K, Verhulst F, Jeppesen P, Jepsen JRM, Vangkilde S, Olsen MH, Hagstrom J, Lonfeldt NN, Plessen KJ. Family-based cognitive behavioural therapy versus family-based relaxation therapy for obsessive-compulsive disorder in children and adolescents: protocol for a randomised clinical trial (the TECTO trial). BMC Psychiatry. 2022 Mar 19;22(1):204. doi: 10.1186/s12888-021-03669-2. PMID 35305587
- See also: Updated systematic review of cognitive behavioural therapy for children and adolescents with obsessive-compulsive disorder — https://www.crd.york.ac.uk/PROSPERO/display_record.php?RecordID=79118